CLINICAL TRIAL: NCT06223165
Title: Evidence-based Sexual and Reproductive Health Intervention Using a Multiphase Optimization Strategy
Brief Title: Optimizing the Floreciendo Sexual and Reproductive Health Workshop for Latina Teens and Female Caregivers: A Pilot
Acronym: Floreciendo
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: Centro Romero (Unknown); Expanded Mental Health Services of Chicago (Unknown); Corazon Community Services (Unknown); Gads Hill Center (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: 2022-0207
Record Dates: First submitted 2024-01-04; First posted 2024-01-25 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Sexual Risk Behavior; Sexually Transmitted Infections; Unplanned Pregnancy
Keywords: Sexual and reproductive health; Latina teens; Mother-daughter intervention
MeSH Terms: conditions — Sexually Transmitted Diseases; Coitus | interventions — Foundations; Condoms; Contraception; Sex; Association

STUDY DESIGN:
Intervention Model Description: We will run a 2 x 2 x 2 pilot factorial experiment. Small groups of Latina teen-female caregiver dyads will be randomized to one of eight conditions. All groups of dyads will receive the constant (i.e., the intervention session focused on foundations in sexual risk prevention). The remaining three intervention components are either delivered (i.e., "on") or not delivered (i.e., "off").
Who Masked: Outcomes Assessor
Masking Description: Recruiters and data collectors will be blind to the intervention condition. Teen-caregiver dyads will not know what intervention condition they are randomized into until they arrive on site for the first workshop session. Key study staff and intervention facilitators will be made aware of the intervention conditions for the purposes of delivering the workshop.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Foundations, Condoms & Contraception, Family Strengthening, and Gender & Relationships (Experimental): This arm receives the constant session (Foundations in Sexual Risk Prevention) and all three other workshop sessions: 1) Condoms & Contraception, 2) Family Strengthening, and 3) Gender & Relationships.
  Interventions: Behavioral: Floreciendo (Foundations, Condoms & Contraception, Family Strengthening, and Gender & Relationships)
- Foundations, Condoms & Contraception, and Family Strengthening (Experimental): This arm receives the constant session (Foundations in Sexual Risk Prevention) and two other workshop sessions: 1) Condoms & Contraception and 2) Family Strengthening.
  Interventions: Behavioral: Floreciendo (Foundations, Condoms & Contraception, and Family Strengthening)
- Foundations, Condoms & Contraception, Gender & Relationships (Experimental): This arm receives the constant session (Foundations in Sexual Risk Prevention) and two other workshop sessions: 1) Condoms & Contraception and 2) Gender & Relationships.
  Interventions: Behavioral: Floreciendo (Foundations, Condoms & Contraception, Gender & Relationships)
- Foundations, Family Strengthening, and Gender & Relationships (Experimental): This arm receives the constant session (Foundations in Sexual Risk Prevention) and two other workshop sessions: 1) Family Strengthening and 2) Gender & Relationships.
  Interventions: Behavioral: Floreciendo (Foundations, Family Strengthening, and Gender & Relationships)
- Foundations and Condoms & Contraception (Experimental): This arm receives the constant session (Foundations in Sexual Risk Prevention) and one other workshop session: Condoms & Contraception.
  Interventions: Behavioral: Floreciendo (Foundations and Condoms & Contraception)
- Foundations and Family Strengthening (Experimental): This arm receives the constant session (Foundations in Sexual Risk Prevention) and one other workshop session: Family Strengthening.
  Interventions: Behavioral: Floreciendo (Foundations and Family Strengthening)
- Foundations and Gender & Partner Relationships (Experimental): This arm receives the constant session (Foundations in Sexual Risk Prevention) and one other workshop session: Gender & Relationships.
  Interventions: Behavioral: Floreciendo (Foundations and Gender & Partner Relationships)
- Foundations (Experimental): This arm receives the constant session (Foundations in Sexual Risk Prevention) only.
  Interventions: Behavioral: Floreciendo (Foundations)

INTERVENTIONS:
Behavioral: Floreciendo (Foundations, Condoms & Contraception, Family Strengthening, and Gender & Relationships) — * Foundations in sexual risk prevention: Covers key topics in sexual and reproductive health and helps participants develop an awareness of sexual behavior risks.
  * Condoms and contraception: Teaches about different forms of condoms and contraception and offers experiential activities on how to use them.
  * Family strengthening: Facilitates learning and practice in how teens and their female caregivers can communicate about sex and addresses family norms and expectations in Latino culture.
  * Gender and relationships: Covers what a healthy relationship looks like and how to recognize intimate partner violence, while discussing how gender and cultural norms in Latino culture influence teens' sexual behavior.
  Arms: Foundations, Condoms & Contraception, Family Strengthening, and Gender & Relationships
Behavioral: Floreciendo (Foundations, Condoms & Contraception, and Family Strengthening) — * Foundations in sexual risk prevention: Covers key topics in sexual and reproductive health and helps participants develop an awareness of sexual behavior risks.
  * Condoms and contraception: Teaches about different forms of condoms and contraception and offers experiential activities on how to use them.
  * Family strengthening: Facilitates learning and practice in how teens and their female caregivers can communicate about sex and addresses family norms and expectations in Latino culture.
  Arms: Foundations, Condoms & Contraception, and Family Strengthening
Behavioral: Floreciendo (Foundations, Condoms & Contraception, Gender & Relationships) — * Foundations in sexual risk prevention: Covers key topics in sexual and reproductive health and helps participants develop an awareness of sexual behavior risks.
  * Condoms and contraception: Teaches about different forms of condoms and contraception and offers experiential activities on how to use them.
  * Gender and relationships: Covers what a healthy relationship looks like and how to recognize intimate partner violence, while discussing how gender and cultural norms in Latino culture influence teens' sexual behavior.
  Arms: Foundations, Condoms & Contraception, Gender & Relationships
Behavioral: Floreciendo (Foundations, Family Strengthening, and Gender & Relationships) — * Foundations in sexual risk prevention: Covers key topics in sexual and reproductive health and helps participants develop an awareness of sexual behavior risks.
  * Family strengthening: Facilitates learning and practice in how teens and their female caregivers can communicate about sex and addresses family norms and expectations in Latino culture.
  * Gender and relationships: Covers what a healthy relationship looks like and how to recognize intimate partner violence, while discussing how gender and cultural norms in Latino culture influence teens' sexual behavior.
  Arms: Foundations, Family Strengthening, and Gender & Relationships
Behavioral: Floreciendo (Foundations and Condoms & Contraception) — * Foundations in sexual risk prevention: Covers key topics in sexual and reproductive health and helps participants develop an awareness of sexual behavior risks.
  * Condoms and contraception: Teaches about different forms of condoms and contraception and offers experiential activities on how to use them.
  Arms: Foundations and Condoms & Contraception
Behavioral: Floreciendo (Foundations and Family Strengthening) — * Foundations in sexual risk prevention: Covers key topics in sexual and reproductive health and helps participants develop an awareness of sexual behavior risks.
  * Family strengthening: Facilitates learning and practice in how teens and their female caregivers can communicate about sex and addresses family norms and expectations in Latino culture.
  Arms: Foundations and Family Strengthening
Behavioral: Floreciendo (Foundations and Gender & Partner Relationships) — * Foundations in sexual risk prevention: Covers key topics in sexual and reproductive health and helps participants develop an awareness of sexual behavior risks.
  * Gender and relationships: Covers what a healthy relationship looks like and how to recognize intimate partner violence, while discussing how gender and cultural norms in Latino culture influence teens' sexual behavior.
  Arms: Foundations and Gender & Partner Relationships
Behavioral: Floreciendo (Foundations) — • Foundations in sexual risk prevention: Covers key topics in sexual and reproductive health and helps participants develop an awareness of sexual behavior risks.
  Arms: Foundations

SUMMARY:
Floreciendo is a sexual and reproductive health workshop for Latina teens (ages 14-18 years) and their female caregivers (e.g., mothers, sisters, grandmothers). This study involves conducting a pilot optimization trial of Floreciendo using the multiphase optimization strategy (MOST) framework. The feasibility of using a 2 x 2 x 2 factorial trial design and the acceptability of the intervention components of Floreciendo will be examined. Effectiveness and implementation outcomes will be explored. This work will be conducted in partnership with community-based organizations in the Chicagoland area.

DETAILED DESCRIPTION:
In the U.S., Latina teens face a disproportionate burden of HIV/AIDS/sexually-transmitted infections (STIs) and other adverse consequences of risky sexual behavior. Parents play a key role in shaping the sexual behavior of their teens as they transition into adulthood. Positive parenting practices-including monitoring, open parent-child communication, and parent-child bonding-have been shown to deter teens' engagement in high-risk behavior. Interventions which engage parents have shown positive effects on youths' sexual health, including among Latinos. Effective Latina mother-daughter sexual health programs are critically needed since Latina mothers are less likely to discuss sexual risk behaviors with their teens than White or Black mothers but are greatly respected as figures of authority in Latine tradition.

This study centers on Floreciendo, a sexual and reproductive health workshop for Latina teens and their female caregivers which was adapted from the evidence-based IMARA (Informed, Motivated, Aware, and Responsible Adolescents and Adults) intervention. Floreciendo is comprised of 4 two-hour sessions, during which teens and caregivers complete separate and joint activities. This study will draw on the multiphase optimization strategy (MOST) framework, an engineering-inspired methodological framework for optimizing an intervention by identifying an intervention package that produces the best expected outcome achievable within key constraints.

The goal of the study is to carry out a pilot optimization trial of Floreciendo using the MOST framework. In partnership with community-based organizations in the Chicagoland area, approximately 92 teen-caregiver dyads (184 participants) will be enrolled. All participants will receive the first workshop session (the constant). In a 2 x 2 x 2 factorial design, small groups of teen-caregiver dyads will be randomized to receive different combinations of the remaining three workshop sessions (the intervention components): 1) condoms & contraception; 2) family strengthening, and 3) gender and relationships. Primary outcomes are: 1) feasibility of using a factorial trial design, and 2) acceptability of the intervention components. We will also explore effectiveness outcomes and implementation outcomes. Data will be collected at baseline and follow-up (roughly 6 months post).

ELIGIBILITY:
Inclusion criteria for teens:

1. Identify as Latina
2. Be 14-18 years old
3. Speak English and/or Spanish
4. Be available and have a female caregiver who is available for the workshop and research activities.
5. Be living with or in daily contact with the female caregiver.

Inclusion criteria for female caregivers:

1. Be the mother or a female caregiver (e.g., aunt, sister, grandmother) of a Latina teen (aged 14-18 years old)
2. Be 19 years old or older
3. Speak English and/or Spanish
4. Be available and have a teen who is available for the workshop and research activities.
5. Be living with or in daily contact with the Latina teen.

Latina teens and female caregivers must agree to participate as a dyad, and teens' refusal will supersede parental consent.

Exclusion Criteria:

Teens and caregivers will be excluded if they are unable to understand the consent/assent process and provide informed consent/assent or if they already received the intervention in a previous phase of the research. Teens may or may not be sexually active; this will not be an exclusion criterium. Information about teens' sexual activity will not be shared with caregivers to reduce consent/assent barriers. If there is more than one eligible adolescent in the family, we will randomly select one to maintain independent observations. Teens or caregivers who become pregnant during the study may continue to participate. Prisoners will be excluded.

Min Age: 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Teens and caregivers must identify as female
Enrollment: 184 (Estimated)
Dates: Start 2024-03-09 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Feasibility of factorial trial design | Through study completion (anticipated 2.5 years)
  Proportion of conditions implemented according to the randomization schedule (benchmark is at least 90%) (primary). We will also measure the proportion of teen-caregiver dyads who complete all sessions specified per their condition (benchmark is at least 80%), and proportion of teen-caregiver dyads who complete baseline assessments (benchmark is at least 80%) and follow-up assessments (benchmark is at least 80%).
Acceptability of intervention components | Immediately after completing the intervention
  Degree of satisfaction with the components of the Floreciendo workshop based on a measure of acceptability adapted from the mental health implementation science tool (mHIST), supplemented with qualitative feedback

OTHER OUTCOMES:
Exploratory primary effectiveness outcome: Sexual risk behavior | Baseline to follow-up
  Proportion of teens who report risky sexual behavior at baseline and follow-up (self-reported using AIDS Risk Behavior Assessment)
Exploratory secondary effectiveness outcome: sexually transmitted infections | Baseline to follow-up
  Proportion of teens with a sexually transmitted infection (STI) at baseline and follow-up.
Exploratory secondary effectiveness outcome: Unplanned pregnancy | Baseline to follow-up
  Proportion of teens with an unplanned pregnancy at baseline and follow-up (self-reported)
Exploratory implementation outcomes | Through study completion (anticipated 2.5 years)
  We will explore feasibility of implementing the Floreciendo intervention, appropriateness, adoption, sustainability, cost, and fidelity.

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Gads Hill Center, Chicago, Illinois
  - Expanded Mental Health Services of Chicago NFP, Chicago, Illinois
  - Centro Romero, Chicago, Illinois
  - Corazon Community Services, Cicero, Illinois

IPD SHARING:
Plan to Share IPD: No